CLINICAL TRIAL: NCT01143519
Title: Effect of SNPs in p53 and p53 Response Elements on the Inflammatory Response to DNA Damage
Brief Title: Study of the Effect of SNPs in p53 and p53 Response Elements on the Inflammatory Response to DNA Damage
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 100134; 10-E-0134
Record Dates: First submitted 2010-06-11; First posted 2010-06-14 (Estimated); Last update posted 2026-01-05 (Actual); Status verified 2025-05-02

CONDITIONS: HIV-1 Seropositive; Inflammation; Cancer; Cardiomyopathy
Keywords: Gene Expression; Apoptosis; Lymphocytes; Environmental Factors; Single Nucleotide Polymorphism; Natural History; Healthy Volunteer; HV
MeSH Terms: conditions — Inflammation; Neoplasms; Cardiomyopathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- FLT1 C-677T: SNP
- MDM2 rs2279744: SNP
- p53 rs1042522: SNP
- RMM1 rs1465952: SNP
- TLR8 rs3761624: SNP

SUMMARY:
Background:

- Research has shown that certain proteins in cells may be linked to higher risks of developing inflammations, tumors, and other medical problems. By examining how the blood cells of healthy volunteers respond to environmental exposures, researchers hope to better understand the relationship of genes, environmental factors, and human diseases.

Objectives:

- To examine how specific genes and proteins in blood cells respond to environmental exposures.

Eligibility:

- Healthy volunteers between 18 and 45 years of age.

Design:

* The study will involve one visit of 45 to 60 minutes.
* Participants will be screened with a brief physical examination and finger stick to determine if they are eligible to donate blood for the study, and will complete a questionnaire about any medications or other drugs (e.g., cigarettes) they may be taking.
* Participants will provide a blood sample for research purposes.

DETAILED DESCRIPTION:
This research study will investigate the role of SNPs in p53 and p53 response elements on the inflammatory response to DNA damage. A total of 200 participants aged 18 years and older carrying one of the five SNPs of interest and wild-type controls will be identified and recruited from the Environmental Polymorphism Registry (EPR). In addition, participants will be recruited based on their health outcomes and SNP associations from the EPR registry to study genotype-phenotype effects on lymphocytes. The EPR is a long-term project to collect and store up to 15,000 DNA samples for use in research studies from individuals in the greater North Carolina Triangle Region.

This observational gene association study will recruit participants on the basis of genotype or phenotype and then observe the lymphocyte response to chemotherapeutic agents and relevant environmental pathogens. The SNPs of interest are p53, as well as four of its downstream target genes including FLT1, MDM2, TLR8 and RRM1. A maximum of 320 mLs of blood will be obtained from each participant during one visit lasting approximately one hour. Cells from the donated blood samples will be examined for their response to exposed environmental stress ex vivo.

The primary objective is to determine the association between five SNPs and p53 target gene expression after exposure to Nutlin or doxorubicin (chemotherapeutic agents) with outcome measured by RT-PCR. The five SNPs are p53 rs1042522, MDM2 rs2279744, FLT1 C-677T, TLR8 rs3761624 and RMM1 rs1465952. The secondary objectives are to: (1) to determine the p53 promoter occupancy measured by ChIP analysis for the following SNPs: FLT1 C-677T, TLR8 rs3761624 and RMM1 rs1465952; (2) to measure apoptosis by Annexin V-PI assay for p53 rs1042522 SNPs; (3) to examine the cell cycle profile analysis (FACS) by cytofluorometry for p53 rs1042522SNPs; and (4) to determine DNA repair using Pulse Field Electrophoresis Gel (TAFE gels) for the following p53 rs1042522SNPs. Furthermore, the association between the SNPs of interest and phenotypic characteristics will be explored using the EPR health and exposure survey to identify significant genotype-phenotype associations in the EPR population. The effect of the associations will be tested on lymphocyte function after exposure to Nutlin or doxorubicin.

We have established that p53 can greatly alter expression of many immune genes including most of the toll-like receptor (TLR) innate immunity genes which are considered important components of antiviral immunity against HIV infection. Given the unique roles of TLR signaling during acute HIV-1 infection and their potential role in chronic inflammation, it is important to elucidate whether TLR polymorphisms contribute to HIV-1 pathogenesis and variability in disease progression.

Recently, we confirmed that p53 can target the TLR8 ssRNA responsive receptor in a single nucleotide polymorphism (SNP)-dependent manner (rs3761624). We have shown in a human study that a SNP within a p53 response element of the TLR8 promoter can strongly influence respiratory syncytial virus (RSV)-associated disease in infants. In addition, there are SNPs in the coding region of p53 that alter the amplitude of signaling attributed to this protein. Projecting these findings to HIV and AIDS, we hypothesize that p53 is a downstream effector that initiates anti-proliferative innate immune responses to viruses and other pathogens, establishing a new role for p53. These novel investigations will provide critical understanding of the role of innate restriction factors in resistance to HIV-1 and disease progression.

Overall, we hope the results of this study lead to discovery of important information regarding the role of SNPs located in p53 and p53 response elements in human disease, potentially identifying new targets for future studies.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Male or female 18 years of age or older
* Participants must be able to understand and provide written informed consent to participate in the study
* Participants must be able to travel to the CRU
* Nonpregnant
* Healthy participants as defined by the International Red Cross guidelines (Healthy means that an individual feels well and can perform normal activities. If the individual has a chronic condition such as diabetes or high blood pressure, healthy also means that they are being treated and the condition is under control).
* Participants with health outcomes identified by genotype-phenotype association studies.
* HIV-1 seropositive under medicament treatment (for HIV P53 and TLR8 groups only) (checked every 6 months at visit)

EXCLUSION CRITERIA:

* Use of immunosuppressants or other immune-modifying drugs [e.g., Rituxan, Humira, Enbrel, Cyclosporin (Neoral, Sandimmune, and SangCya), Azathioprine (Imuran)], Monoclonal antibodies [e.g., infliximab (Remicade)] (for healthy controls only)
* Chronic use of systemic, inhaled steroids
* Current or use of prescription strength topical corticosteroids within the last 7days
* History of cancer, including skin cancer (for healthy controls only)
* History of chemotherapy or radiation treatment (for healthy controls only)
* Confirmed or suspected immunosuppressive or immunodeficient condition (for healthy controls only)
* Hepatitis B/C-positive status (checked every 6 months at visit)
* Body weight < 50 kg (<110 lbs)
* If blood donation exceeds 200ml:

  --Hematocrit <34% for women or <36% for men, or >56% for either gender
* Temperature > 37.6 C; blood pressure < 90/50 mm Hg or blood pressure >160/100 mm Hg; pulse rate < 50 or > 100 beats/minute
* Blood or plasma donation that will cause the participant to exceed 550ml of blood in the last 8 weeks
* HIV1 donors with opportunistic infections:

  * Candidiasis of bronchi, trachea, esophagus, or lungs
  * Invasive cervical cancer
  * Coccidioidomycosis
  * Cryptococcosis
  * Cryptosporidiosis, chronic intestinal (greater than 1 month's duration)
  * Cytomegalovirus disease (particularly CMV retinitis)
  * Encephalopathy, HIV-related
  * Herpes simplex: chronic ulcer(s) (greater than 1 month's duration); or bronchitis, pneumonitis, or esophagitis
  * Histoplasmosis
  * Isosporiasis, chronic intestinal (greater than 1 month's duration)
  * Kaposi's sarcoma
  * Lymphoma, multiple forms
  * Mycobacterium avium complex
  * Tuberculosis
  * Pneumocystis carinii pneumonia
  * Pneumonia, recurrent
  * Progressive multifocal leukoencephalopathy
  * Salmonella septicemia, recurrent
  * Toxoplasmosis of brain
  * Wasting syndrome due to HIV

    * HIV and hepatitis results will be confidentially obtained. Testing will be contracted to an external certified laboratory. Results will be available only to the study team, with the few caveats that follow:

All positive HIV, hepatitis B, and hepatitis C results that are unexpected (i.e. participant is not currently enrolled in the EPR as an HIV-1 seropositive under medicament treatment) will be promptly communicated to the donor by the study doctor/PI or the CRU Director. The participant will be referred to their physician and/or to the N.C. Department of Health for confirmatory testing and counseling. As explained in detail in the attached Supplement describing N.C. State Department of Health code will be followed. The state code mandates reporting of positive results along with the participant s name and identifying information to the N.C. Department of Public Health. Upon contracting with the testing laboratory, clarification will be obtained and documented as to whether the contracted laboratory or the study MD will be responsible for reporting positive results to the state to avoid duplication of reporting. Upon receipt of the test results, the N.C. Department of Health will contact the participant to inform them of the positive result, how to find care, how to avoid infecting others, how the newly diagnosed HIV and/or hepatitis infection is reported, and the importance of informing their partners at possible risk because of their HIV and/or hepatitis infection. If the HIV, hepatitis B, and hepatitis C results are negative, the participant will be not be notified. However, the participant may contact the research study nurse for their results.

HIV and hepatitis B/C test results, non-reactive and reactive, will be documented confidentially by the PI or study coordinator in the subject s file, and kept in a locked file cabinet in the CRU Medical Records Room. In order to document the reporting procedure and the time associated with the reporting process, a document has been created and placed in the study specific manual (Hepatitis B/C and HIV Notification Process for Reactive Results Form).

-Healthy control participants carrying SNPs TLR8 and FLT1 who are currently taking hormonal contraception (e.g. oral contraceptives, IUDs with hormones, contraceptive patches) or hormone replacement therapy will be excluded from the study unless the participant has been off of the hormone treatment for 1 month or longer.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants at the age of 18 years and older carrying one of the following SNPs: p53 rs1042522, MDM2 rs2279744, FLT1 C-677T, TLR8 rs3761624 and RMM1 rs1465952 in the p53 promoter region or in p53 target gene RE regions and wild-type controls will be identified from the Environmental Polymorphism Registry (EPR).
Sampling Method: Non-Probability Sample
Enrollment: 178 (Actual)
Dates: Start 2012-05-21 (Actual)

PRIMARY OUTCOMES:
p53 target gene expression | analysis on blood drawn at visit
  The primary endpoint of this study is p53 target gene expression measured by RTPCR for the following five SNPs: p53 rs1042522, MDM2 rs2279744, FLT1 C-677T, TLR8 rs3761624 and RMM1 rs1465952.

SECONDARY OUTCOMES:
p53 promoter occupancy | analysis on blood drawn at visit
  Measured by ChIP analysis for the following SNPs: FLT1 C-677T, TLR8 rs3761624 and RMM1 rs1465952.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Menendez Rendon, Ph.D., Principal Investigator — National Institute of Environmental Health Sciences (NIEHS)
Locations (1):
- NIEHS Clinical Research Unit (CRU), Research Triangle Park, North Carolina, United States

REFERENCES:
- [Background] Bond GL, Hu W, Bond EE, Robins H, Lutzker SG, Arva NC, Bargonetti J, Bartel F, Taubert H, Wuerl P, Onel K, Yip L, Hwang SJ, Strong LC, Lozano G, Levine AJ. A single nucleotide polymorphism in the MDM2 promoter attenuates the p53 tumor suppressor pathway and accelerates tumor formation in humans. Cell. 2004 Nov 24;119(5):591-602. doi: 10.1016/j.cell.2004.11.022. PMID 15550242
- [Background] Menendez D, Inga A, Resnick MA. The expanding universe of p53 targets. Nat Rev Cancer. 2009 Oct;9(10):724-37. doi: 10.1038/nrc2730. PMID 19776742
- [Background] Murphy ME. Polymorphic variants in the p53 pathway. Cell Death Differ. 2006 Jun;13(6):916-20. doi: 10.1038/sj.cdd.4401907. No abstract available. PMID 16557270
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2010-E-0134.html